CLINICAL TRIAL: NCT05665881
Title: Effects of Vasopressors on Cerebral Hemodynamics in Patients With Carotid Endarterectomy Under General Anesthesia(TCD Part): a Randomized Controlled Study
Brief Title: Effects of Vasopressors on Cerebral Hemodynamics in Patients With Carotid Endarterectomy (TCD Part)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Ruquan Han, Professor & Director, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: wxy20220513
Record Dates: First submitted 2022-05-26; First posted 2022-12-27 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Carotid Endarterectomy
Keywords: carotid endarterectomy; ephedrine; phenylephrine; norepinephrine; cerebrovascular circulation; cerebral blood flow hemodynamics
MeSH Terms: interventions — Ephedrine; Phenylephrine; Norepinephrine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: This study could not be blinded to the treating anesthesiologists. However, blinding was maintained for the patients and the assessors of outcome indicators. Postoperative follow-up was performed by a specially trained physician who did not have access to any information about the patients' cases and subgroups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ephedrine (Experimental): Ephedrine group: receive ephedrine (configured concentration 2 mg/mL). The individualized blood pressure control target was a 10% increase in baseline blood pressure, and the target blood pressure value was used as the basis for adjusting the dosing or pumping rate.
  Interventions: Drug: Ephedrine
- Phenylephrine (Experimental): Phenylephrine group: receive intravenous infusion of phenylephrine (configured concentration 0.1 mg/mL) The individualized blood pressure control target was a 10% increase in baseline blood pressure, and the target blood pressure value was used as the basis for adjusting the dosing or pumping rate.
  Interventions: Drug: Phenylephrine
- norepinephrine (Experimental): norepinephrine group: intravenous infusion of norepinephrine (configured concentration of 6 μg/ml).The individualized blood pressure control target was a 10% increase in baseline blood pressure, and the target blood pressure value was used as the basis for adjusting the dosing or pumping rate.
  Interventions: Drug: Norepinephrine

INTERVENTIONS:
Drug: Ephedrine — vasopressor
  Arms: Ephedrine
Drug: Phenylephrine — vasopressor
  Arms: Phenylephrine
Drug: Norepinephrine — vasopressor
  Arms: norepinephrine

SUMMARY:
This study was a single-center, exploratory, randomized controlled trial. First, the effects of ephedrine, phenylephrine, or norepinephrine on cerebral blood flow hemodynamics in patients undergoing carotid endarterectomy were evaluated using TCD techniques to investigate the specific mechanisms of the three vasopressors on cerebral blood flow and oxygen metabolism in brain tissues.

DETAILED DESCRIPTION:
Carotid endarterectomy is a procedure used to remove plaque from the common and internal carotid arteries and improve cerebral perfusion. Clinical studies have demonstrated the effectiveness of this procedure in both symptomatic and asymptomatic patients. intraoperative circulatory management challenges in carotid endarterectomy include the following: ① the incidence of preoperative combined coronary artery disease, hypertension and diabetes mellitus is relatively high in patients undergoing carotid endarterectomy, and there is a pathological basis for systemic vascular injury, increasing the risk of perioperative cardiovascular and cerebrovascular complications, such as myocardial ischemia and stroke. ② During the CEA procedure, the common carotid artery, internal carotid artery and external carotid artery and the superior thyroid artery need to be blocked respectively, the source of blood supply to the cerebral hemisphere on the operated side is reduced and depends only on the Willis circle supply. ③ Carotid sinus pressure receptor pull stimulation causes circulatory fluctuations. During CEA, a relatively high arterial pressure is required to provide adequate cerebral perfusion. However, achieving this target blood pressure level intraoperatively can be challenging due to given conditions, the presence of induction drugs and anesthetics. Therefore, it is particularly important to maintain cerebral hemodynamic stability and ensure tissue perfusion with intraoperative use of vasopressors.

The purpose of this study was to evaluate the effects of ephedrine, phenylephrine, or norepinephrine on cerebral blood flow hemodynamics in CEA patients using TCD techniques to investigate the specific mechanisms of the three boosting agents on cerebral blood flow and oxygen metabolism in brain tissues.

ELIGIBILITY:
Inclusion Criteria:

1. age 40-80 years.
2. elective carotid endarterectomy.
3. Signed informed consent

Exclusion Criteria:

1. American Society of Anesthesiologists physical status classification (ASA) IV - VI.
2. renal failure (estimated glomerular filtration rate less than 60 ml/min.m2).
3. cardiac arrhythmias.
4. Allergy to ephedrine, phenylephrine or norepinephrine, gadobutrol.
5. patients with preoperative TCD suggesting poor temporal window signal.
6. patients with severe carotid artery stenosis with no flow signal detected by TCD
7. Patients with tandem lesions of carotid artery stenosis

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-01-07 (Actual); Primary Completion 2024-09-24 (Actual); Study Completion 2024-09-24 (Actual)

PRIMARY OUTCOMES:
Changes in middle cerebral artery blood velocity | 10 minutes after entering the operating room; 10 minutes after intubation ;5 minutes after administration of vasopressors
  This outcome is measured by transcranial doppler ultrasound.

SECONDARY OUTCOMES:
Changes in regional oxygen saturation index | 10 minutes after entering the operating room; 10 minutes after intubation ;5 minutes after administration of vasopressors
  This outcome is measured by Near Infrared Spectroscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided